CLINICAL TRIAL: NCT06127108
Title: Multi-center Clinical Evaluation of the Panbio™ COVID-19/Flu A&B Panel
Brief Title: Clinical Evaluation of the Panbio™ COVID-19/Flu A&B Panel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2319801
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Influenza A; Influenza B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Study staff will collect two (2) anterior nasal swabs from each Participant.
  One anterior nasal swab will be collected by a study staff member and tested immediately on the Panbio™ COVID-19/Flu A&B Panel by an untrained test operator. The other anterior nasal swab will be eluted in VTM within 10 minutes of sample collection. The swab will be rotated vigorously in the VTM, and the swab head will be left in the VTM, by snapping the shaft or clipping the base of the swab if necessary. VTM samples will be stored, handled and tested with comparator assays according to the manufacturers' product instructions. VTM specimens can be stored for up to 48 hours at 2-8°C. If delivery and processing of samples exceeds specified time periods, specimens should be transported in dry ice and once in laboratory frozen at -70°C or colder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Nasal sampling/Testing (professional use) (Experimental): Operator or delegated study staff will collect one anterior nasal swab sample from both nostrils. The collected anterior nasal swab will the tested with the Panbio™ COVID-19/Flu A&B Panel by the operator at the study site in a near patient testing setting (e.g. GP center or hospital clinic). After the anterior nasal swab is collected, the operator or delegated study staff will collect one anterior nasal swab from both nostrils of the subject for RT-PCR testing. VTM samples will be shipped daily to the central lab for testing with the RT-PCR protocols for Flu A, Flu B and SARS-CoV-2.
  Interventions: Diagnostic Test: Panbio™

INTERVENTIONS:
Diagnostic Test: Panbio™ — The Panbio™ COVID-19/Flu A&B Panel is a visual lateral flow in vitro immunoassay for the qualitative detection of the nucleocapsid protein antigen to SARS-CoV-2, Influenza A, and Influenza B in anterior nasal swab samples from individuals with symptoms and suspected of COVID-19 or Flu infection by their healthcare provider.
  Other Names: Panbio™ COVID-19/Flu A&B Panel

SUMMARY:
The study is designed as a prospective, multicentric, clinical study to investigate the positive percent agreement (PPA) and negative percent agreement (NPA) of the Panbio™ COVID-19/Flu A&B Panel using anterior nasal swab specimens tested directly, relative to the comparator methods, Roche cobas® SARS-CoV-2 (K231306) and Quidel Lyra® Influenza A+B Assay(K230236) (RT-PCR) in symptomatic patients suspected of respiratory viral infection by a healthcare provider.

DETAILED DESCRIPTION:
Approximately 2,000 symptomatic Participants to achieve at least 80 COVID-19 PCR confirmed positives, 80 Flu A PCR confirmed positives, 80 Flu B PCR confirmed positives, and 500 COVID-19 and Influenza PCR-confirmed negatives.

Site staff will collect two (2) anterior nasal swabs from each Participant from whom informed consent has been obtained. Participants ages two (2) years and older meeting eligibility criteria will be enrolled.

One anterior nasal swab will be immediately eluted in an extraction buffer tube and tested with the Panbio™ COVID-19/Flu A&B Panel. If immediate testing is not possible, the swab specimen can be kept in an extraction buffer tube filled with extraction buffer at room temperature (59-86°F /15-30 °C) for up to one (1) hour prior to testing.

The other anterior nasal swab will be rotated vigorously in VTM, and the swab head will be left in the VTM, by snapping the shaft or clipping the base of the swab if necessary.

Anterior nasal swab sample collection will be as follows:

With the swab designated for Panbio testing, use gentle rotation to push the swab into the right nostril until resistance is met at the level of the turbinates (less than one inch into the nostril). Rotate the swab several times against the nasal wall then slowly remove from the nostril. Using the swab designated for PCR testing, repeat sample collection in the left nostril.

With the swab designated for PCR testing, use gentle rotation to push the swab into the right nostril until resistance is met at the level of the turbinates (less than one inch into the nostril). Rotate the swab several times against the nasal wall then slowly remove from the nostril. Using the swab designated for Panbio testing, repeat sample collection in the left nostril.

The VTM samples will be stored, handled, and tested with comparator assays according to the manufacturers' product instructions. VTM specimens can be stored for up to 48 hours at 2-8°C. If delivery and processing of samples exceeds specified time periods, specimens should be transported in dry ice and once in laboratory frozen at -70°C or colder.

Swab eluate samples containing the swab head in VTM will be tested at the central laboratory with the Roche cobas® SARS-CoV-2 (K231306) and Quidel Lyra® Influenza A+B Assay (K230236) per product instructions. All discordant samples (i.e., samples with the Roche cobas® SARS-CoV-2 (K231306) or Quidel Lyra® Influenza A+B Assay (K230236) results that conflict with the Panbio™ COVID-19/Flu A&B Panel results) will be evaluated with the Hologic SARS-CoV-2/Flu A/B/RSV Assay (Panther Fusion® System) for information only. Samples may also be tested for viral culture.

Note: For the purposes of the COVID-19 method comparison, Roche cobas® SARS-CoV-2 results will be interpreted per the package insert. Roche cobas® SARS-CoV-2 results where the ORF1a/b (Target 2) is Negative or Invalid and the E-Gene (Target 3) is Positive are considered Presumptive Positive for COVID-19. These samples will be further evaluated with the Hologic SARS-CoV-2/Flu A/B/RSV Assay (Panther Fusion® System).

Each Participant's demographic data, inclusion/exclusion data, days of symptom onset, comparator results, Panbio™ COVID-19/Flu A&B Panel results and other data elements will be recorded as detailed in Section 10 of this document. Defined Participant data will be recorded on source documentation and entered into an Electronic Data Capture (EDC) system. Panbio™ results and the comparator method results will not be provided to study Participants. Panbio™ COVID-19/Flu A&B Panel test operators will be blinded to a Participant's standard of care COVID-19 and/or Flu test results.

ELIGIBILITY:
Inclusion Criteria:

* Participant is suspected of acute viral respiratory infection by a healthcare professional, and
* Participant is age two (2) years or older, and
* Participant is within seven (7) days of symptom onset, and
* Participant is experiencing two or more of the following symptoms:
* Fever of >100.0°F/ 37.8°C
* Cough
* Fatigue
* New loss of taste or smell
* Congestion or runny nose
* Shortness of breath or difficulty breathing
* Sore throat
* Muscle or body aches
* Headache
* Nausea or vomiting
* Diarrhea

Exclusion Criteria:

* Participant is currently enrolled in a study to evaluate an investigational drug or experimental treatment
* Participants with an active nosebleed
* Participant has undergone a nasal wash or nasal aspirate procedure on day of enrollment
* Participant has received a nasal spray or mist Influenza vaccine (i.e. FluMist) within the last 30 days
* Participant has tested positive for COVID-19 within the last 45 days (excluding test results received after current onset of symptoms)
* Participant has received antiviral medications for Influenza (Amantadine, Rimantadine, Ribavirin, Oseltamivir, Zanamivir) in the previous 45 days
* Participant has received medication or treatment for COVID-19 infection in the last 45 days (including antivirals, convalescent plasma therapy, monoclonal antibody treatment (mAb), Remdesivir, long-acting antibody (LAAB) treatment (Evusheld)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA | "up to 24 months"
  1. Primary Outcome: The primary objective of this study is to demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA) of the Panbio™ COVID-19/Flu A&B Panel using anterior nasal swab specimens tested directly, relative to the comparator methods, the Roche cobas® SARS-CoV-2 (K231306) and Quidel Lyra® Influenza A+B Assay (K230236) (RT-PCR) in symptomatic patients suspected of respiratory viral infection by a healthcare provider. Samples may also be tested for viral culture.

SECONDARY OUTCOMES:
Demonstrate the accuracy of the Panbio™ COVID-19/Flu A&B Panel in the hands of untrained users by a usability questionnaire. | "Up to 24 months"
  Secondary Outcome:
  The secondary objective of this study is to demonstrate the accuracy of the Panbio™ COVID-19/Flu A&B Panel in the hands of untrained users, which are "intended users" in a point of care (POC) Clinical Laboratory Improvement Amendments of 1988 (CLIA) moderate, high or waived complexity test environment.
  Each test operator will be given a user evaluation questionnaire once to assess the usability of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Pediatrics, Vienna, Virginia, United States

IPD SHARING:
Plan to Share IPD: No